CLINICAL TRIAL: NCT04868357
Title: Efficacy of Self-administered Hypnosis for the Complementary Management of Anxiety and Dyspnea During Pulmonary Rehabilitation: A 2-armed Randomized Controlled Trial
Brief Title: Hypnosis for the Management of Anxiety and Breathlessness During a Pulmonary Rehabilitation Program
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier de Bligny (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: HYPNOBPCO_2
Record Dates: First submitted 2021-04-23; First posted 2021-04-30 (Actual); Last update posted 2026-01-05 (Actual); Status verified 2025-12

CONDITIONS: COPD; Dyspnea; Anxiety
Keywords: COPD; Dyspnea; Anxiety; Depression; Hypnosis
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Dyspnea; Anxiety Disorders; Depression | interventions — Hypnosis

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hypnosis (Experimental): Delivered twice during the 4-week PRP program (weeks 1,3). It consists of 45-minute sessions of group hypnosis. It includes 1 hypnotic induction, multiple suggestions of relaxation and a feeling of air entering the lungs, and a closing exercise. The intervention includes a prescription to use these exercises freely throughout the PRP, as a tool for self-managing discomfort and inducing calmness. This arm is structured following the classic format of didactic hypnosis interventions, were patients discover the exercise by doing it, and receive keys to be able to recreate the hypnotic state on their own.
  Interventions: Behavioral: Hypnosis
- Relaxation (Active Comparator): Delivered twice during the 4-week PRP program (weeks 1,3). It consists of 45-minute sessions of group dynamic relaxation. It includes 1 exercise to liberate tension, 3 exercises to increase proprioception and calmness, and 3 exercises for calming and regulating the breath. The intervention includes a prescription to use these exercises freely throughout the PRP, as a tool for self-managing discomfort and inducing calmness.
  1. Provides additional care that motivates the patients to participate in the control group.
  2. Allows the controlling of number of group interventions accross arms (2).
  3. Allows to control for motivation, as both arms are introduced identically: the benefits and interest of using self-relaxation techniques for complementary care in anxiety and anxiety-related dyspnea are underscored.
  4. It allows the disentanglement of hypnosis and relaxation effects . This was crucial, inasmuch as hypnosis too includes physical relaxation and breathing exercises.
  Interventions: Behavioral: Relaxation

INTERVENTIONS:
Behavioral: Hypnosis — Two 45-minute group sessions in which patients experience hypnosis and learn how to use it for the self-management of anxiety and anxiety-related dyspnea. First session is introductory. Second session addresses concerns that patients may have identified after using self-hypnosis. Both sessions include group hypnosis exercises. Both sessions are to be administered in an identical manner, and require the same motor and communication responses from the patient (i.e., concentrate on the practitioner's voice, eye closure, relaxation, nodding). Patients are asked to concentrate in nature-themed metaphors and hypnotic suggestions of pure air entering their lungs. Both sessions end with a round of questions, instructions and motivation to use self-hypnosis throughout the duration of the PRP and beyond.
  Arms: Hypnosis
Behavioral: Relaxation — Two 45-minute group sessions in which patients experience dynamic relaxation and learn how to use it for the self-management of anxiety and anxiety-related dyspnea. Both sessions include group relaxation exercises. Both sessions are to be administered in an identical manner, and require the same motor and communication responses from the patient (i.e., concentrate on the practitioner's voice, stretching, breathing exercises, nodding). Both sessions end with a round of questions, instructions and motivation to use relaxation throughout the duration of the PRP and beyond.
  Arms: Relaxation

SUMMARY:
Patients with chronic obstructive pulmonary disease (COPD) are prone to breathlessness, chest tightness and other anxiety-inducing symptoms. Medical therapy for the condition focus on improving these symptoms and preventing exacerbations. However, as the disease progresses, pharmacological therapies become less and less effective. Patients with advanced COPD often feel less benefit from the treatment in terms of relief from their symptoms and relief from anxiety about their breathing. Hypnosis is known to induce immediate changes in how a person thinks and experiences their body. These changes can break vicious cycles of anxiety. Hypnosis has already been used successfully people with breathing problems to reduce anxiety and improve breathing. This trial aims to investigate the effect of hypnosis as a complementary technique for the self-management of breathlessness and anxiety during a Pulmonary Rehabilitation Program (PRP). As a secondary measure, the investigators aim to uncover whether the use of self-hypnosis remains useful during the three months following the PRP, after discharge from hospital.

DETAILED DESCRIPTION:
Chronic Obstructive Pulmonary Disease (COPD) is a highly prevalent and debilitating respiratory condition characterized by chronic airflow limitation, increased respiratory rate, dyspnea and other persistent respiratory symptoms. Growing evidence associates dyspnea to a higher risk of experiencing anxiety, depression and suicidality. In stable COPD, the prevalence of clinical depression ranges between 10% and 42%, and prevalence of anxiety between 10% and 19%. A definitive causal link between these conditions can be hard to establish: symptoms of depression, anxiety and COPD frequently overlap. However, the management of these comorbidities in tandem with COPD is of central importance, as evidence has shown that the alleviation of anxiety symptoms can improve COPD prognosis and increase rehabilitation completion rates. The American Thoracic Society consensus statements on COPD have acknowledged that medical and pharmacological treatments, when used alone, are of limited efficacy for the relief of dyspnea and anxiety in people with advanced COPD. Psychological and complementary management of COPD has been strongly encouraged, and evidence in its favor has been promising so far. Furthermore, because of the interactions between anxiety, depression and chronic dyspnea, it has been proposed that proper assessment and comprehensive management of COPD could constitute a Human Rights matter, and psychological care together with well-informed choice of intervention should be a fundamental complement to standard treatment. The GOLD initiative for COPD acknowledges the benefits from cognitive behavioral therapy and mind-body interventions (mindfulness-based therapy, yoga, relaxation and others) for managing anxiety and depression in patients with COPD. However, despite its numerous advantages (rapid effect, easy and fast implementation, virtually no effort required on behalf of the patient) the efficacy of hypnosis for COPD complementary anxiety management remains scarcely evaluated.

In HYPNOBPCO_1, the investigators found that COPD-related anxiety responded positively to hypnosis (vs sham). The investigators found that a scripted, 15-minute hypnosis session improved anxiety levels, respiratory rate and arterial oxygen saturation. In particular, anxiety as assessed through STAI-6 scores (State-Trait Anxiety Inventory - 6 items), decreased a mean percentage of (Standard Deviation [SD]) -23.8% [18.4] after the hypnosis session (χ2=28, Degrees of Freedom=1, P < 0.0001, Bayes Factor = 1212), equivalent to an 11.2 [9.2] point reduction in STAI-6 score. The difference in anxiety improvement between hypnosis and sham was itself significant (χ2=8, DF=1, P < 0.01, BF = 5.5).

HYPNOBPCO_2 seeks to answer some of the queries that were beyond the scope of its predecessor. The investigators intend to evaluate the efficacy of hypnosis as complementary care during a Pulmonary Rehabilitation Program (PRP). This long-duration protocol will focus on the complementary management and self-management of chronic anxiety in COPD patients through hypnosis. The investigators shall evaluate if the positive effects of hypnosis withstand repeated use, persist when hypnosis is self-administered, and estimate their general impact on psychological and physiological outcomes of COPD patients admitted for a PRP in the PRP conducted by the Centre Hospitalier de Bligny (CHB).

**Baseline Characteristics**

Information other than clinical endpoints of interest is included, to control for confounds and ensure both arms remain comparable:

Age: in years. Sex: male/female CI: Charlson Comorbidity Index; BMI: body mass index; FEV1: forced expiratory volume in 1s; FVC: forced vital capacity; FEV1/FVC: Tiffeneau score; BODE Index: BODE composite score for gravity assessment; mMRC score: Modified Research Council Questionnaire; PaO2: oxygen partial arterial pressure; PaCO2: carbon dioxide partial arterial pressure; GOLD: Global Initiative for Obstructive Lung Disease 2006 and 2011 criteria (1-4/A-D); Oxygenotherapy: Long term (LTO) or ambulatory. HADS score: Hospital Anxiety and Depression scale score. 6MWD: 6-minute walk distance test; CAT: COPD assessment test; MDP: Multidimensional Dyspnea Profile. STAI-6 score: State-trait anxiety inventory - 6 item version. Anxiety-related psychoactive drug intake: dosage/frequency Morphine use: dosage/frequency **Data dictionary** Descriptions of each variable are provided. This dictionary bridges the English terminology with the standard French lexicon used by the CHB throughout PRP and standard hospitalization.

6MWT: 6 minute Walk Test BMI: Body Mass Index BPCO: Bronchopneumopathie Chronique Obstructive (equivalent to COPD) CAT: COPD Assessment Test CHB: Centre Hospitalier de Bligny (Bligny Hospital Center) COPD: Chronic Obstructive Pulmonary Disease (equivalent to BPCO) VEMS: Volume expiratoire maximal/seconde (equivalent to FEV1) VEMS/CV: Volume expiratoire maximal/seconde/Capacité Vitale (equivalent to Tiffeneau score) FR: Fréquence Respiratoire (eq. to Respiratory Rate) CV/CPT: Capacité Vitale/Capacité Pulmonaire Totale (eq. to FVC over total lung capacity).

GOLD: Global Initiative for Chronic Obstructive Lung Disease HAD: Hospital Anxiety and Depression Scale MDP: Multidimensional Dyspnea Profile mMRC: modified Medical Research Council scale PRP: Programme de Réhabilitation Pulmonaire (eq. to Pulmonary Rehabilitation Program) SpO2: Saturation d'Oxygène - saturation pulsée (eq. pulsated oxygen saturation) STAI-6: State-trait Anxiety Inventory - 6 Item version VO2peak: Peak Oxygen Uptake VSRQ: Visual Simplified Respiratory Questionnaire WRpeak: Peak Work Rate CCI: Charlson comorbidity index.

Results will be reported in English.

**Quality assurance plan** Data validation and registry procedures will be monitored and validated by the Quality Control Agent(s) selected by the sponsor. The expert(s) will be independent from the trial.

**Data checks** Data will be entered into a secured digital registry, following a predefined format. Data forms were developed under the supervision of CHB's care providers and chest physicians, who assessed data collection feasibility. Consistency across data fields will be checked at the beginning and end of each PRP.

**Source data verification** Digital data will proceed directly from CHB's patient records, and from paper forms containing all outcomes not already comprised by standard health monitoring during PRP. Digital records will be compared to paper records prior being send for data analysis, to ensure validity.

**Standard Operating Procedures** Operating procedures have been agreed upon prior trial registration. Care providers in the CHB will approach PRP patients and advertise the trial. Patients interested in the trial will be provided with a detailed leaflet explaining the trial's layout and goal (partially masking hypothesis to prevent motivation biases). Patients who decide to participate will be screened for inclusion criteria. Those who follow inclusion criteria will be asked to sign an informed consent and be told that they will be included in either the Hypnosis Arm or the Dynamic Relaxation Arm. At that time, a unique random 3-digit numerical ID will be assigned to each patient to ensure participant anonymity throughout the trial. Importantly, the CHB can only conduct one PRP at the time, and patients participating of said PRP are in contact with each other during group activities (under strict safety protocols). Hence, it was deemed impractical to conduct both arms of the study simultaneously during a single PRP instance. Main concerns included patients sharing self-hypnosis and relaxation techniques with each other across arms, and the generation of motivation biases or attrition out of wanting to switch groups. Since it is fundamental that the trial is conducted in conditions close to a normal CHB's PRP, separation of the participants or prevention of group activities were discarded. Hence, all patients participating of a given PRP instance will be inscribed in either the Active Control or Treatment arm of the trial. To ensure a balanced randomization under these circumstances, a hospital representative will produce an amount of sealed envelopes equal to the total amount of PRPs that will compose the entire trial. Half of the envelopes will assign "Active Control" as intervention, and the other half will assign "Treatment". Before the beginning of each PRP, one envelope will be drawn at chance. This envelope will determine which intervention will take place during that PRP. Neither the care-givers, the patients or the investigators will have any influence or prior knowledge on which envelop is drawn, nor will they have the possibility to refuse drawing outcome. Data will be collected through paper forms by care providers involved in the trial. Digitalization will be performed on anonymized data exclusively. Arms will remain masked to investigators in charge of analyzing outcome changes. Special adverse effect forms have been made available to care providers, and a pipeline with the sponsor to report adverse events and enact a potential emergency stop of the trial have been established.

**Sample size assessment** Results from HYPNOBPCO_1 indicate that a sample of N=20 are sufficient to detect an instant, transient effect of hypnosis over anxiety. However, HYPNOBPCO_2 targets lasting effects of hypnosis over anxiety, influence of repeated use, self-administration, and impact on PRP concurrent outcomes. Thus, larger samples may be needed. Preliminary effect-size analyses for primary outcomes will be conducted once the threshold of 20 patients is achieved. These values will then be used in an a-priori simulation-based power analysis (power >= 80%, alpha=0.05) to estimate desired sample size. Recruitment will continue until the target established by this prior analysis is reached. If required sample size exceeds 100 participants (50 patients per arm), continuation of the trial will be subjected to deliberation (due to material limitations of the CHB). If the sponsor and the investigators agree, the trial will be pursued beyond 100 participants and the record will be amended.

**Plan for missing data** The investigators will conduct our statistical analyses using mixed-effect models. This will allow us to retain participants even if some data instances remain unavailable, or are considered uninterpretable because of data inconsistencies or out-of-range results. However, participants presenting half or more instances of missing data will be excluded.

**Statistical analysis plan** The investigators will performed data analysis using R. The investigators will consider the differences between baseline and outcome scores. The investigators will also contrast these differences across interventions (Hypnosis vs Relaxation). Indicators will be modeled by implementing linear (mixed) models, with a random intercept per participant. A hierarchical modeling approach will allow us to account for individual participant differences, and for imbalances in sample size across factors and levels. Significance tests will be computed by means of likelihood ratio tests that compare our models to simpler models, in which the relevant predictor will be removed. ANOVA tables will be computed through Analysis of Deviance (Type II Wald χ2 test), and post hoc pairwise comparisons through Tukey contrasts of least-squares means, setting a 95 % CI. Findings will be considered statistically significant when P value <0.05.

To prove lack of effect the investigators will calculate an approximation of the Bayes Factor from the Bayesian Information Criterion, for the saturated and null models implicated in the contrast (BIC approximation to BF, so that BF = exp ((BICnull-BICfull)/2)). The BF will account for the strength of evidence in favor of the full model, meaning BF < 1 equal virtual lack of effect, and BF > 2 equal a strong, noteworthy effect.

ELIGIBILITY:
Inclusion Criteria:

* Aged > 30.
* Affiliated to a Social Security scheme or beneficiary of such a scheme.
* Absence of cognitive disease questioning the validity of patient reported outcomes
* Ability to give free, informed consent.
* Adult patients with severe COPD, dyspnea ; with distension.
* Hospitalized at the CHB.
* Predicted FEV1 and FEV/FVC percentages consistent with severe COPD according to GOLD standards.
* Modified Research Council Questionnaire ≥2
* Exposure to tobbacco >= 10 packs/yrs.

Exclusion Criteria:

* Pregnancy
* Known severe cardiac insufficiency.
* Known severe pulmonary arterial hypertension.
* Evolutive-cancer diagnosis.
* Significant cognitive impairment, hypercapnic encephalopathy or confusional syndrome.
* Deafness.
* Anemia ≤ 8g/dL.
* Psychotic pathology.

Ages: 30 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 133 (Actual)
Dates: Start 2021-09-27 (Actual); Primary Completion 2024-04-19 (Actual); Study Completion 2024-04-19 (Actual)

PRIMARY OUTCOMES:
Change in anxiety scores | Baseline (inclusion in PRP, Week 1). Week 2. Week 3. Week 4 (PRP completion). After finishing the PRP, once a month for 3 months.
  Anxiety, as determined by the State-Trait Anxiety Inventory (6 item version, STAI-6). This scale rates anxiety with a score between 20 and 80 points. The cutoff score for a clinical anxiety diagnosis is 39 points. Lower scores mean lower anxiety levels.
Change in anxiety & depression scores | Baseline (inclusion in PRP, Week 1). Week 4 (PRP completion).
  Anxiety, as determined by the Hospital Anxiety and Depression inventory (HADS). This scale rates anxiety and depression tendencies with a score between 0 and 21. The cutoff score for a clinical mild anxiety diagnosis is 8-10 points. Lower scores mean lower anxiety and depression levels.
Change in anxiety and quality of life scores | Baseline (inclusion in PRP, Week 1). Week 4 (PRP completion).
  Anxiety and quality of life as measured by the Multidimensional Dyspnea Profile. The MDP consists of 11 items divided into three domains (discomfort breathing by intensity, discomfort breathing by description, anxiety and distress coming from breathing difficulties). In all domains, intensity is rated from 0 (negligible) to 10 (worst possible condition). In the second domain in particular, the respondent selects between five descriptors the one that better represents their breathing discomfort, and then rates its intensity. Lower levels mean less discomfort and better quality of life.

SECONDARY OUTCOMES:
6-minute walking test | Baseline (inclusion in PRP, Week 1). Week 4 (PRP completion).
  This exercise test measures the distance the patient can walk quickly on a flat, hard surface in six minutes. It reflects the patient's ability to perform daily physical activities.
COPD Assesment Test (CAT) | Baseline (inclusion in PRP, Week 1). Week 4 (PRP completion). After finishing the PRP, once a month for 3 months.
  Full assessment of the COPD Assesment Test.
Re-hospitalisation rate | After finishing the PRP, once a month for 3 months.
  Inquiring wether the patient has been hospitalized again after the PRP, in connection to dyspnea, exacerbation, or anxiety. To be obtained through monthly telephonic interviews.
Use of self-hypnosis techniques | A measure completed by the patient throughout the PRP up to 4 weeks. Then once a month after finishing the PRP for 3 months.
  A questionnaire developed at the CHB asking simply whether patients used hypnosis to manage their anxiety and breathlessness, how many times a week, and whether they felt satisfied with hypnosis effects.
Action Plan | Once a month after finishing the PRP, for 3 months.
  Occurrences of use of an action plan including corticoids and/or antibiotics after PRP.
  Delivered at discharge, detailed explanations on the use of this plan having been done during dedicated workshops, as part of the PRP.

OTHER OUTCOMES:
Smoking status. | Baseline (inclusion in PRP, Week 1). Week 4 (PRP completion). Once a month after finishing the PRP, for 3 months.
  An exploratory variable. Monitoring how many cigarettes do patients smoke a day.
Psychoactive drug intake | Baseline (inclusion in PRP, Week 1). Week 4 (PRP completion). Once a month after finishing the PRP, for 3 months.
  An exploratory variable. Anxiety-related psychoactive drug intake (dosage/frequency)

CONTACTS AND LOCATIONS:
Overall Officials: François Larue, MD, Study Director — Centre Hospitalier de Bligny
Locations (1):
- Centre Hospitalier de Bligny, Briis-sous-Forges, Briis-sous-Forges, France

IPD SHARING:
Plan to Share IPD: Yes
The anonymized data will be available for free, upon request to the Centre Hospitalier de Bligny. The Centre Hospitalier de Bligny will only share the data to inquirers capable of respecting the conditions established by the Commission Nationale de l'Informatique et des Libertés for data protection (CNIL, https://www.cnil.fr/). Please address any questions to the corresponding author at hernan.anllo@cri-paris.org.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data will be available upon request for the 10 years after the publication of the study
Access Criteria: The Centre Hospitalier de Bligny will only share the data to inquirers capable of respecting the conditions established by the Commission Nationale de l'Informatique et des Libertés for data protection (CNIL, https://www.cnil.fr/).

REFERENCES:
- [Background] Vogelmeier CF, Criner GJ, Martinez FJ, Anzueto A, Barnes PJ, Bourbeau J, Celli BR, Chen R, Decramer M, Fabbri LM, Frith P, Halpin DM, Lopez Varela MV, Nishimura M, Roche N, Rodriguez-Roisin R, Sin DD, Singh D, Stockley R, Vestbo J, Wedzicha JA, Agusti A. Global Strategy for the Diagnosis, Management and Prevention of Chronic Obstructive Lung Disease 2017 Report: GOLD Executive Summary. Respirology. 2017 Apr;22(3):575-601. doi: 10.1111/resp.13012. Epub 2017 Mar 7. PMID 28150362
- [Background] Han MK, Muellerova H, Curran-Everett D, Dransfield MT, Washko GR, Regan EA, Bowler RP, Beaty TH, Hokanson JE, Lynch DA, Jones PW, Anzueto A, Martinez FJ, Crapo JD, Silverman EK, Make BJ. GOLD 2011 disease severity classification in COPDGene: a prospective cohort study. Lancet Respir Med. 2013 Mar;1(1):43-50. doi: 10.1016/S2213-2600(12)70044-9. Epub 2012 Sep 3. PMID 24321803
- [Background] Pumar MI, Gray CR, Walsh JR, Yang IA, Rolls TA, Ward DL. Anxiety and depression-Important psychological comorbidities of COPD. J Thorac Dis. 2014 Nov;6(11):1615-31. doi: 10.3978/j.issn.2072-1439.2014.09.28. PMID 25478202
- [Background] Hegerl U, Mergl R. Depression and suicidality in COPD: understandable reaction or independent disorders? Eur Respir J. 2014 Sep;44(3):734-43. doi: 10.1183/09031936.00193213. Epub 2014 May 29. PMID 24876171
- [Background] Kellner R, Samet J, Pathak D. Dyspnea, anxiety, and depression in chronic respiratory impairment. Gen Hosp Psychiatry. 1992 Jan;14(1):20-8. doi: 10.1016/0163-8343(92)90022-3. PMID 1730397
- [Background] Maurer J, Rebbapragada V, Borson S, Goldstein R, Kunik ME, Yohannes AM, Hanania NA; ACCP Workshop Panel on Anxiety and Depression in COPD. Anxiety and depression in COPD: current understanding, unanswered questions, and research needs. Chest. 2008 Oct;134(4 Suppl):43S-56S. doi: 10.1378/chest.08-0342. PMID 18842932
- [Background] Di Marco F, Verga M, Reggente M, Maria Casanova F, Santus P, Blasi F, Allegra L, Centanni S. Anxiety and depression in COPD patients: The roles of gender and disease severity. Respir Med. 2006 Oct;100(10):1767-74. doi: 10.1016/j.rmed.2006.01.026. Epub 2006 Mar 13. PMID 16531031
- [Background] Cafarella PA, Effing TW, Usmani ZA, Frith PA. Treatments for anxiety and depression in patients with chronic obstructive pulmonary disease: a literature review. Respirology. 2012 May;17(4):627-38. doi: 10.1111/j.1440-1843.2012.02148.x. PMID 22309179
- [Background] Parshall MB, Schwartzstein RM, Adams L, Banzett RB, Manning HL, Bourbeau J, Calverley PM, Gift AG, Harver A, Lareau SC, Mahler DA, Meek PM, O'Donnell DE; American Thoracic Society Committee on Dyspnea. An official American Thoracic Society statement: update on the mechanisms, assessment, and management of dyspnea. Am J Respir Crit Care Med. 2012 Feb 15;185(4):435-52. doi: 10.1164/rccm.201111-2042ST. PMID 22336677
- [Background] Basoglu M. Effective management of breathlessness: a review of potential human rights issues. Eur Respir J. 2017 May 25;49(5):1602099. doi: 10.1183/13993003.02099-2016. Print 2017 May. No abstract available. PMID 28546267
- [Background] Tselebis A, Pachi A, Ilias I, Kosmas E, Bratis D, Moussas G, Tzanakis N. Strategies to improve anxiety and depression in patients with COPD: a mental health perspective. Neuropsychiatr Dis Treat. 2016 Feb 9;12:297-328. doi: 10.2147/NDT.S79354. eCollection 2016. PMID 26929625
- [Background] Smith SM, Sonego S, Ketcheson L, Larson JL. A review of the effectiveness of psychological interventions used for anxiety and depression in chronic obstructive pulmonary disease. BMJ Open Respir Res. 2014 Nov 3;1(1):e000042. doi: 10.1136/bmjresp-2014-000042. eCollection 2014. PMID 25478188
- [Background] Hynninen MJ, Bjerke N, Pallesen S, Bakke PS, Nordhus IH. A randomized controlled trial of cognitive behavioral therapy for anxiety and depression in COPD. Respir Med. 2010 Jul;104(7):986-94. doi: 10.1016/j.rmed.2010.02.020. Epub 2010 Mar 25. PMID 20346640
- [Background] Lolak S, Connors GL, Sheridan MJ, Wise TN. Effects of progressive muscle relaxation training on anxiety and depression in patients enrolled in an outpatient pulmonary rehabilitation program. Psychother Psychosom. 2008;77(2):119-25. doi: 10.1159/000112889. Epub 2008 Jan 25. PMID 18230945
- [Background] Volpato E, Banfi P, Rogers SM, Pagnini F. Relaxation Techniques for People with Chronic Obstructive Pulmonary Disease: A Systematic Review and a Meta-Analysis. Evid Based Complement Alternat Med. 2015;2015:628365. doi: 10.1155/2015/628365. Epub 2015 Aug 3. PMID 26339268
- [Background] Vickers A, Zollman C. ABC of complementary medicine. Hypnosis and relaxation therapies. BMJ. 1999 Nov 20;319(7221):1346-9. doi: 10.1136/bmj.319.7221.1346. No abstract available. PMID 10567143
- [Background] Montgomery GH, Sucala M, Baum T, Schnur JB. Hypnosis for Symptom Control in Cancer Patients at the End-of-Life: A Systematic Review. Int J Clin Exp Hypn. 2017 Jul-Sep;65(3):296-307. doi: 10.1080/00207144.2017.1314728. PMID 28506144
- [Background] Anllo H, Herer B, Delignieres A, Bocahu Y, Segundo I, Mach Alingrin V, Gilbert M, Larue F. Hypnosis for the Management of Anxiety and Dyspnea in COPD: A Randomized, Sham-Controlled Crossover Trial. Int J Chron Obstruct Pulmon Dis. 2020 Oct 22;15:2609-2620. doi: 10.2147/COPD.S267019. eCollection 2020. PMID 33122899